CLINICAL TRIAL: NCT02054364
Title: Feasibility of Combining Family and Cognitive Therapy to Prevent Chronic Anorexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, James Dale Lock, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH101281 (NIH); Grant Funding Number (NIH) (Other Grant/Funding Number: SPO#109319)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorder; Anorexia Nervosa; Eating Disorder Not Otherwise Specified; Maudsley; Family-Based Therapy; FBT; Family Therapy; Cognitive Remediation Therapy; CRT
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FBT and CRT (Experimental): Family-Based Treatment combined with Cognitive Remediation Therapy (15 sessions of each)
  Interventions: Behavioral: FBT and CRT
- FBT and art therapy (Experimental): Family-Based Treatment combined with art therapy (15 sessions of each)
  Interventions: Behavioral: FBT and art therapy

INTERVENTIONS:
Behavioral: FBT and CRT
  Other Names: Family-Based Treatment (FBT) combined with Cognitive Remediation Therapy (CRT)
  Arms: FBT and CRT
Behavioral: FBT and art therapy
  Other Names: Family-Based Treatment (FBT) combined with art therapy.
  Arms: FBT and art therapy

SUMMARY:
This study aims to investigate the feasibility of combining Cognitive Remediation Therapy (CRT) with Family Based Treatment (FBT) for future use in a randomized clinical trial to reduce the risk of adolescents developing persistent Anorexia Nervosa. Participants will be randomly assigned to one of two groups: one group will receive FBT and CRT, and the other group will receive FBT and art therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for anorexia nervosa Lives with at least one English-speaking parent who is willing to participate Medically Stable Endorses obsessions/compulsions Adequate transportation to clinic Proficient at speaking, reading, and writing English

Exclusion Criteria:

* Previous FBT or CRT for AN Medical Instability Medical condition that may affect eating or weight

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Full remission from AN (%MBW>95) | End of Treatment (6 months)
  Weight restoration to at least 95% of Median body weight (calculated by height, weight, gender, and age)

CONTACTS AND LOCATIONS:
Overall Officials: James Lock, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- See also: Program information — http://edresearch.stanford.edu